CLINICAL TRIAL: NCT01479985
Title: Randomized Clinical Trial of a Computerized Contraceptive Decision Aid
Brief Title: Computerized Contraceptive Decision Aid
Acronym: CDM RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SFP5-8 -201112047
Record Dates: First submitted 2011-11-17; First posted 2011-11-28 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Contraception; Decision Making; Satisfaction; Evaluation
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDM Tool (Experimental): participants will be randomized to completing the CDM tool
  Interventions: Other: CDM Tool
- Control (No Intervention): Participants will fill out a computer survey similar to CDM tool without the decisive factors and computer print out

INTERVENTIONS:
Other: CDM Tool — Participants will be required to complete the CDM tool and receive a tailored print out of their contraceptive options based on survey answers
  Arms: CDM Tool

SUMMARY:
The purpose of this study is to conduct a randomized clinical trial of a web-based contraceptive decision aid compared to routine contraceptive counseling to evaluate the effect of the contraceptive decision aid on the contraceptive method selected by the participant.

The investigators primary hypothesis is that women utilizing a computerized Contraceptive Decision Aid (CDA) will be more likely to choose highly effective contraception than women who undergo standard clinical contraceptive counseling.

DETAILED DESCRIPTION:
Our primary specific aim is to test the CDA by conducting a randomized clinical trial comparing the CDA to routine contraceptive counseling. Our primary outcome of interest will be selection of highly effective contraception including the intrauterine device (IUD), the implant, and injectable contraception compared to all other reversible contraceptive methods.

We will also complete the following secondary specific aims:

1. We will use the validated Decisional Conflict Scale to measure decisional conflict pre- and post-intervention and compare the change in decisional conflict score in women randomized to the CDA to women undergoing routine counseling.
2. We will also evaluate satisfaction with contraceptive counseling and contraceptive continuation and satisfaction at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45 years old
* At risk for unintended pregnancy and seeking reversible contraception at Center of Advanced Medicine or Washington University Resident's Clinic
* Willing and able to complete Contraceptive Decision Making tool
* English speaking

Exclusion Criteria:

* Have had a hysterectomy, bilateral oophorectomy, have undergone female sterilization
* Unable to give informed consent secondary to language barrier or cognitive limitation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tessa E Madden, MD, MPH, Principal Investigator — Washington University School of Medicine

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CDM Tool | Control
Started | 167 | 86
Baseline Survey | 166 | 85
Completed | 161 | 80
Not Completed | 6 | 6
Not completed — Tablet malfunction, no data saved | 1 | 1
Not completed — No decisional conflict scale responses | 0 | 2
Not completed — No post-visit survey | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDM Tool | Control | Total
Number analyzed (Participants) | 166 | 85 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (6.2) | 28.4 (6.2) | 28.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 85 | 251
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 62 | 23 | 85
  White | 84 | 55 | 139
  Other | 20 | 7 | 27
Region of Enrollment [Number; unit: participants]
  United States | 166 | 85 | 251

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict Scale Score
Description: Pre-Visit, Post-Visit and change in Decisional Conflict Scale (DCS) Score between Post-Visit (immediately following visit) and Pre-Visit (immediately prior to visit). The Decisional Conflict Scale scores range from 0 to 100; 0 represents no decisional conflict and 100 represents high decisional conflict.
Time Frame: Pre-Visit and Post-Visit (same day)
Population: 8 subjects did not complete the post-visit survey, so a post-visit DCS score and change in DCS score could not be calculated
Measure: Median (Full Range); unit: score on a scale
Arm/Group | CDM Tool | Control
Number analyzed (Participants) | 166 | 83
score on a scale
  Pre-Visit Score | 15 [0 to 80] | 10 [0 to 85]
  Post-Visit Score: number analyzed (Participants) | 161 | 80
  Post-Visit Score | 0 [0 to 70] | 0 [0 to 35]
  Change in Score: number analyzed (Participants) | 161 | 80
  Change in Score | -10 [-80 to 25] | -10 [-60 to 5]

2. Secondary Outcome: Contraceptive Method Chosen
Description: Contraceptive method chosen at end of visit with healthcare provider as reported on the post-visit survey
Time Frame: Post-visit (immediately after visit)
Measure: Count of Participants; unit: Participants
Arm/Group | CDM Tool | Control
Number analyzed (Participants) | 161 | 80
Participants
  LNG-IUS | 45 | 21
  Copper IUD | 9 | 3
  Implant | 9 | 6
  DMPA | 19 | 4
  Pills | 57 | 29
  Contraceptive patch | 1 | 0
  Vaginal ring | 8 | 5
  Sterilization | 0 | 3
  Condoms | 7 | 4
  Other | 1 | 3
  No method/undecided | 5 | 2

ADVERSE EVENTS:
Arm/Group | CDM Tool | Control
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/86
Other Adverse Events (participants affected / at risk) | 0/167 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No